CLINICAL TRIAL: NCT00508326
Title: Phase I Study of Paclitaxel Administered by Hepatic Artery Infusion to Patients With Advanced Cancer and Dominant Liver Involvement
Brief Title: Paclitaxel Administered by HAI to Patients With Advanced Cancer and Dominant Liver Involvement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0092
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Solid Tumor; Liver Metastasis; Hepatic Artery Infusion; Liver; Paclitaxel; Taxol
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HAI Paclitaxel (Experimental): Paclitaxel via Hepatic Artery Infusion (HAI)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Starting dose 150 mg/m^2 HAI once every 4 weeks
  Other Names: Taxol

SUMMARY:
The goal of this clinical research study is find the highest tolerated dose of paclitaxel that can be given directly into the liver of patients with advanced cancer involving the liver. Researchers also want to collect descriptive information on any effects the drug may have on tumor tissue.

DETAILED DESCRIPTION:
Paclitaxel is designed to work by blocking the mechanisms of cell division in cancer cells, causing them to die.

Before you can start on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have a complete medical history and physical exam, including measurement of height, weight, and vital signs (blood pressure, temperature, breathing rate, and heart rate). You will have a neurological evaluation evaluating your strength and nerve function. You will be asked to report how a pinprick or a thin brush feel when applied to your skin. About 2 tablespoons of blood and some urine samples will be collected for routine tests. Women who are able to have children must have a negative urine pregnancy test.

If you are eligible to take part in this study, you will begin taking study drugs in cycles of 28 days. You will be hospitalized to receive your chemotherapy. The night of the hospital admission, you will receive fluids (normal saline) in your veins to help decrease the risk of kidney side effects from the chemotherapy. The morning after your admission to the hospital, you will be taken to the interventional radiology suite, and a catheter (a thin plastic tube) will be placed in your groin area and advanced to the liver. You must be on bedrest the entire time that the catheter is in place. After the procedure, you will go to Nuclear Medicine, and a test called "flow study" will be carried out to confirm the right position of the catheter. After your return to the room, the nurses will start the chemotherapy. You will receive paclitaxel nonstop over 24 hours through the catheter (a thin plastic tube) into the artery that carries blood to your liver. You will repeat this procedure once every month.

The catheter will be carefully taped so that it can not move and to prevent it from coming out while you are receiving chemotherapy. You will be asked to lie flat on your back while the treatment takes place. In some cases, the catheter will be removed immediately after your chemotherapy infusions is complete. In some cases, the catheter will remain in longer. You will be on bedrest until the catheter is removed. When the catheter is pulled, pressure will be applied to the groin for 15 minutes. The catheter will be removed by someone experienced in the procedure. The catheter will be placed and removed for each cycle of chemotherapy. Blood (about 2 teaspoons) will be drawn for blood counts and liver function tests, before each dose, to be sure researchers are safely giving you the paclitaxel.

You will be seen by a doctor or advanced practitioner every day while you are in the hospital. You will be hospitalized for about 3-5 days until recovery from all immediate chemotherapy-related side effects. The charges of your hospitalization will be billed to you or your insurance carrier.

You will continue to receive the chemotherapy once every 28 days, unless the disease gets worse or intolerable side effects occur. Every 2 months and at the end of your participation in this study, you will have scans to see if your tumors are growing or shrinking and blood work (about 3 teaspoons) will be performed for safety tests. These tests can be performed at your doctor's office and the results faxed to the study doctor at M. D. Anderson.

In addition, you will be asked to call the research nurse in charge of this study at 713-745-1042 to report on your health status every week for 30 days after the last dose of the drug or until you start a new course of therapy.

This is an investigational study. The chemotherapy you will be given is FDA approved. The cost of being on these medications will be billed to you or your insurance company. About 59 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed diagnosis of advanced malignancy and liver involvement as dominant site of metastasis.
2. Performance status ECOG < or = 2 (Requires occasional assistance but is able to care for own needs).
3. Adequate renal function (serum creatinine < 2.0 mg/dL).
4. Adequate hepatic function (Total bilirubin < 2.0 mg/dL; ALT </= 5 times upper normal reference value).
5. Bone marrow function (ANC >or =1.5 cells/mcL; PLT > or = 100,000 cells/mcL).
6. At least three weeks from previous therapy and complete recovery from all associated acute toxicities.
7. Ability to fully read, comprehend, and sign informed consent forms.
8. All females in childbearing age must have a negative urine or serum HCG test unless prior hysterectomy or menopause. Women of childbearing potential and men must use effective birth control.
9. Patients should be refractory to standard chemotherapy or have no conventional therapy that produces a CR rate of at least 10% or an increase in survival of at least three months.
10. Patients of both genders, 13 year-old or older.

Exclusion Criteria:

1. Clinical or radiographic evidence of ascites.
2. Pregnant or breastfeeding females.
3. Hypersensitivity to paclitaxel compounds.
4. History of severe hypersensitivity reactions to products containing polyoxyethylated castor oil or Cremophor.
5. Inability to complete informed consent process and adhere to protocol treatment plan and follow-up requirements.
6. Untreatable bleeding diathesis.
7. Portal vein thrombosis.
8. Peripheral neuropathy > Grade 1 according to NCI CTC v.3.0: sensory alteration not interfering with function).
9. Untreated (radiation therapy, chemotherapy, surgery or a combination of modalities) brain metastasis.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of Monthly Cytotoxic Intraarterial Hepatic Paclitaxel | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia M. Tsimberidou, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org